CLINICAL TRIAL: NCT02024711
Title: EYEFILL® C.-US Viscoelastic Clinical Investigational Protocol- For Institutional Review Boards / Ethical Review Committees and Clinical Investigators
Brief Title: EYEFILL® C. -US Viscoelastic Clinical Investigation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Collaborators: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EYE-C-7.00
Record Dates: First submitted 2013-12-27; First posted 2013-12-31 (Estimated); Results first posted 2020-09-04 (Actual); Last update posted 2020-09-04 (Actual); Status verified 2020-09

CONDITIONS: Cataract
Keywords: Cataract; Intraocular Lens; IOL; Aphakia
MeSH Terms: conditions — Cataract; Aphakia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- EYEFILL® C.-US Viscoelastic (Experimental): EYEFILL ® C.-US is designed for use during cataract extraction and intraocular lens implantation surgery to protect the corneal endothelium, and other intraocular tissues and to manipulate tissues during these anterior chamber ocular surgeries.
  Interventions: Device: EYEFILL® C.-US Viscoelastic
- Healon® Viscoelastic (CONTROL) (Active Comparator): Healon® is designed for use during cataract extraction and intraocular lens implantation surgery to protect the corneal endothelium, and other intraocular tissues and to manipulate tissues during these anterior chamber ocular surgeries.
  Interventions: Device: Healon® Viscoelastic (CONTROL)

INTERVENTIONS:
Device: EYEFILL® C.-US Viscoelastic — EYEFILL ® C.-US is designed for use during cataract extraction and intraocular lens implantation surgery to protect the corneal endothelium, and other intraocular tissues and to manipulate tissues during these anterior chamber ocular surgeries.
  Arms: EYEFILL® C.-US Viscoelastic
Device: Healon® Viscoelastic (CONTROL) — Healon® is designed for use during cataract extraction and intraocular lens implantation surgery to protect the corneal endothelium, and other intraocular tissues and to manipulate tissues during these anterior chamber ocular surgeries.
  Arms: Healon® Viscoelastic (CONTROL)

SUMMARY:
The purpose of this multicenter, prospective, randomized clinical study is to determine the safety and effectiveness of the EYEFILL® C.-US Viscoelastic in patients undergoing cataract extraction and intraocular lens (IOL) implantation surgery.

EYEFILL® C.-US Viscoelastic is designed to create and maintain space, to protect the corneal endothelium and other intraocular tissues, and to manipulate tissues during surgery.

EYEFILL® C.-US Viscoelastic may also be used to coat intraocular lenses and instruments during cataract extraction and intraocular lens insertion.

ELIGIBILITY:
Inclusion Criteria:

* Any race
* Older than 21 years
* Cataract requiring cataract extraction in at least 1 eye
* Clear intraocular media other than cataract
* Able to provide written informed consent
* Able and willing to comply with required follow-up schedule
* Competent to understand the procedure and the actions asked of him/her as a research subject

Exclusion Criteria:

* Monocular
* Ocular infection
* History of glaucoma, Ocular Hypertension (IOP > 21 mmHg) likely to require IOP lowering medications, ocular condition requiring IOP lowering medication, condition preventing reliable Goldmann applanation tonometry, known steroid responder
* Previous intraocular surgery in the operative eye
* Previous serious corneal disease or known endothelial cell loss / damage (in operative eye)
* History of chronic or recurrent inflammatory eye disease (in operative eye)
* Evidence of retinal vascular disease (in operative eye)
* Uncontrolled diabetes or proliferative diabetic retinopathy
* Acute or chronic disease or illness that would increase the operative risk
* Allergy to anesthetics or other postoperative medications
* Known hypersensitivity to sodium hyaluronate or other components in viscoelastic
* Patient in any other clinical trial within the 30 days prior to the start of the study

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 262 (Actual)
Dates: Start 2013-12; Primary Completion 2014-12-17 (Actual); Study Completion 2014-12-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donald R Sanders, MD, PhD, Study Director — Center for Clinical Research
Locations (8):
- United States (8):
  - Barnet Dulaney Perkins Eye Center, Phoenix, Arizona
  - Shasta Eye Medical Group, Redding, California
  - Argus Research at Cape Coral Eye Center, Cape Coral, Florida
  - Eye Centers of Florida, Fort Myers, Florida
  - Newsom Eye and Laser Center, Sebring, Florida
  - Great Lakes Eye Care, Saint Joseph, Michigan
  - Silverstein Eye Centers, Kansas City, Missouri
  - Comprehensive Eye Care, Washington, Missouri

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | EYEFILL® C.-US Viscoelastic | Healon® Viscoelastic (CONTROL)
Started | 130 | 132
Completed | 129 | 128
Not Completed | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | EYEFILL® C.-US Viscoelastic | Healon® Viscoelastic (CONTROL) | Total
Number analyzed (Participants) | 130 | 132 | 262
Age, Continuous [Mean (Full Range); unit: years] | 69.4 [39 to 83] | 68.7 [36 to 86] | 69.0 [36 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75 | 78 | 153
  Male | 55 | 54 | 109

OUTCOME MEASURES:

1. Primary Outcome: Mean Percent Cell Change (Preservation of Endothelium)
Description: Preservation of endothelium was assessed by specular microscope photographs to determine endothelial cell density.
Time Frame: Baseline, 3 months
Population: Participants with endothelial cell density recorded at baseline and 3 months are included in the population.
Measure: Mean (Standard Deviation); unit: percent cell change
Arm/Group | EYEFILL® C.-US Viscoelastic | Healon® Viscoelastic (CONTROL)
Number analyzed (Participants) | 130 | 127
percent cell change | -10.05 (15.06) | -10.13 (15.92)

2. Secondary Outcome: Percentage of Participants With Intraocular Pressure (IOP) Spikes >/= 30 mmHg Any Postoperative Visit
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | EYEFILL® C.-US Viscoelastic | Healon® Viscoelastic (CONTROL)
Number analyzed (Participants) | 130 | 132
Participants | 24 | 20

3. Secondary Outcome: Percentage of Participants With Anterior Chamber Inflammation
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | EYEFILL® C.-US Viscoelastic | Healon® Viscoelastic (CONTROL)
Number analyzed (Participants) | 130 | 132
Participants
  Day 1 | 2 | 4
  Day 7 | 2 | 3
  Day 30 | 4 | 3
  Day 90 | 0 | 0

4. Secondary Outcome: Percentage of Participants With Device-related Adverse Events Any Visit
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | EYEFILL® C.-US Viscoelastic | Healon® Viscoelastic (CONTROL)
Number analyzed (Participants) | 130 | 132
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 3 months
Description: Adverse events were not coded. Therefore, source vocabulary is not applicable.
Arm/Group | EYEFILL® C.-US Viscoelastic | Healon® Viscoelastic (CONTROL)
Serious Adverse Events (participants affected / at risk) | 1/130 | 2/132
Other Adverse Events (participants affected / at risk) | 69/130 | 72/132
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | EYEFILL® C.-US Viscoelastic (N=130) | Healon® Viscoelastic (CONTROL) (N=132)
Total colon blockage (Gastrointestinal disorders) | 0 | 1
Death due to undiagnosed cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Blood clot (Vascular disorders) | 1 | 0
Hematoma (Vascular disorders) | 1 | 0
Anemia (Blood and lymphatic system disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | EYEFILL® C.-US Viscoelastic (N=130) | Healon® Viscoelastic (CONTROL) (N=132)
Corneal stromal edema (Eye disorders) | 41 | 41
Posterior capsular opacity (Eye disorders) | 20 | 19
Macular degeration (Eye disorders) | 8 | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Contact sponsor directly for details.